CLINICAL TRIAL: NCT01869296
Title: The Effect of Endoscopy Water Pump Flow Rates on Successful Unsedated Colonoscopy by Water Immersion Method: a Randomized Controlled Trial
Brief Title: The Effect of Endoscope Water Pump Flow Rates on Successful Unsedated Colonoscopy by Water Immersion Method: a Randomized Controlled Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gadjah Mada University (Other)
Responsible Party: Principal Investigator, PUTUT BAYUPURNAMA, MD, Internist-Gastroenterologist, Gadjah Mada University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: PB-02-CWUGM
Record Dates: First submitted 2013-05-26; First posted 2013-06-05 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: Effect of Endoscope Water Pump Flow Rates
Keywords: unsedated; water immersion colonoscopy; endoscope water pump flow rates

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- higher flow rates endoscope pump (Active Comparator): higher flow rates endoscope water pump : 10.4 ml/sec
  Interventions: Procedure: higher flow rates
- lower flow rates endoscope water pump (Experimental): lower flow rates endoscope water pump : 1.7 ml/sec
  Interventions: Procedure: lower flow rates

INTERVENTIONS:
Procedure: higher flow rates — higher flow rates endoscope pump water immersion colonoscopy : 10.4 ml/sec
  Arms: higher flow rates endoscope pump
Procedure: lower flow rates — lower flow rates endoscope pump water immersion colonoscopy : 1.7 ml/sec
  Arms: lower flow rates endoscope water pump

SUMMARY:
The purpose of this study is to compare the cecal intubation rate between two endoscopy water pump with different flow rates (1.7 ml/sec vs 10.4 ml/sec) in water immersion colonoscopy examination in unsedated patients undergoing diagnostic colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Adult > 18 years old with indication for colonoscopy, such as chronic diarrhea, chronic constipation, hematochezia, chronic lower abdominal pain, positive fecal occult blood test, and other change of bowel habit symptoms indicative of need for diagnostic colonoscopy examination

Exclusion Criteria:

* Patients refuse to participate, patient with obstructive lesion in the colon distal of the cecum, patients with experienced of colon resection, hemodynamically unstable, severe cardiac disorders (such as acute myocardial infarction, unstable angina, malignant arrhythmia, and moderate to severe congestive heart failure), patients with fecal obstruction (whatever the causes) so that impossible to pass the scope through the obstructed segment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2013-05; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
cecal intubation rate | 1.5 years

SECONDARY OUTCOMES:
Cecal intubation time | 1.5 years
Abdominal discomfort score | 1.5 years
Willingness to repeat | 1.5 years
Causes of unsuccessful | 1.5 years
Abdominal compression | 1.5 years
Position change | 1.5 years
Diagnostic lesions | 1.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Putut Bayupurnama, MD, Principal Investigator — Div of Gastroenterology and Hepatology, Dept of Internal Medicine,Fac of Medicine, Gadjah Mada University/Dr.Sardjito General Hospital,Yogyakarta,Indonesia
Locations (1):
- Dr. Sardjito General Hospital, Yogyakarta, Special Region of Yogyakarta, Indonesia

REFERENCES:
- [Derived] Bayupurnama P, Ratnasari N, Indrarti F, Triwikatmani C, Maduseno S, Nurdjanah S, Leung FW. Endoscope-connected water pump with high flow rates improves the unsedated colonoscopy performance by water immersion method. Clin Exp Gastroenterol. 2018 Jan 12;11:13-18. doi: 10.2147/CEG.S152669. eCollection 2018. PMID 29391819